CLINICAL TRIAL: NCT01371617
Title: A Phase 2 Study of IPI-926 in Patients With Myelofibrosis
Brief Title: A Phase 2 Study With IPI-926 in Patients With Myelofibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Infinity Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPI-926-08
Record Dates: First submitted 2011-06-09; First posted 2011-06-13 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2012-11

CONDITIONS: Primary Myelofibrosis; Fibrosis, Bone Marrow
Keywords: IPI-926; 926; Myelofibrosis; Hedgehog; Infinity Pharmaceuticals; Post Essential thrombocythemia; Post Polycythemia vera
MeSH Terms: conditions — Primary Myelofibrosis | interventions — IPI-926

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IPI-926 (Experimental): Single Arm, Phase 2 trial evaluating the safety and efficacy of IPI-926 in patients with myelofibrosis
  Interventions: Drug: IPI-926

INTERVENTIONS:
Drug: IPI-926 — Single Arm study of oral IPI-926 at 160 mg, 130 mg or 110 mg daily, until progressive disease or intolerability to study treatments or withdrawal of ICF
  Other Names: Hedgehog Inhibitor; Hedgehog Pathway Inhibitor

SUMMARY:
The purpose of this study is to determine the safety and efficacy of IPI-926 in patients with myelofibrosis (MF) (primary myelofibrosis [PMF], post-polycythemia vera myelofibrosis [post-PV MF], or post-essential thrombocythemia myelofibrosis [post-ET MF]).

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age at the time of signing the ICF.
* Voluntarily sign an ICF.
* Pathologically confirmed PMF or post ET/PV MF as per the WHO diagnostic criteria (note that it must include at least Grade 1 marrow fibrosis, see Appendix 3) with intermediate-1, intermediate -2, or high risk disease according to the IWG prognostic scoring system (see Appendix 4). If patients have low risk disease, then they must have symptomatic splenomegaly that is ≥ 10 cm below left costal margin by physical exam.
* ECOG performance of 0-2.
* Life expectancy of at least 3 months.
* Recovery to Grade 1 or baseline of any toxicities due to prior systemic treatments, excluding alopecia.
* If a woman, be of non-child bearing potential or, for women of child-bearing potential (WCBP) (defined as a sexually mature woman who has not undergone surgical sterilization or who has not been naturally post-menopausal for at least 24 consecutive months for women ≤55 years; for women >55 years 12 consecutive months), must have a negative serum or urine pregnancy test result within 2 weeks of first dose of study drug.
* All WCBP and all sexually active male patients must agree to use adequate methods of birth control throughout the study. Adequate methods of contraception include use of oral contraceptives with an additional barrier method, double barrier methods (diaphragm with spermicidal gel or condoms with contraceptive foam), Depo-Provera, partner vasectomy, and total abstinence.
* Ability to adhere to the study visit schedule and all protocol requirements.

Exclusion Criteria:

* Prior treatment with any inhibitor of the hedgehog pathway (e.g. GDC-0449).
* Received any treatment for myelofibrosis within 2 weeks of study entry.
* Other invasive malignancies diagnosed within the last 3 years, except non-melanoma skin cancer and localized cured prostate and cervical cancer.
* Inadequate hepatic function defined by:
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >2.5 x upper limit of normal (ULN).
* Direct bilirubin >1.5 x ULN.
* Cirrhotic liver disease, ongoing alcohol abuse, or known chronic active or acute hepatitis.
* Inadequate renal function defined by serum creatinine >2 x ULN.
* History of stroke, unstable angina, myocardial infarction, or ventricular arrhythmia requiring medication or mechanical control within the last 6 months.
* Presence of active infection or systemic use of antibiotics within 72 hours of treatment.
* Significant co-morbid condition or disease, which in the judgment of the Investigator, would place the patient at undue risk or interfere with the study.
* Known human immunodeficiency virus (HIV) positivity.
* Known hypersensitivity to IPI-926, or any of the excipients in IPI-926 capsules.
* Pregnant or lactating women.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
To determine the overall response rate of IPI-926, defined as clinical improvement (CI); partial remission (PR); and complete remission (CR), according to the International working group (IWG) criteria in patients with Myelofibrosis | At least 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Srdan Verstovsek, M.D.; Ph.D, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - Arizona Mayo Clinic, Scottsdale, Arizona
  - Stanford University School of Medicine, Division of Hematology, Palo Alto, California
  - The University of Texas MD Anderson Cancer Center, Houston, Texas